CLINICAL TRIAL: NCT01429519
Title: A PRELIMINARY OPEN CLINICAL STUDY, TO ASSESS THE SAFETY AND EFFICACY OF RPh201 APPLIED TOPICALLY FOR THE TREATMENT OF HARD TO HEAL CHRONIC ULCERATED WOUNDS
Brief Title: Efficacy of RPh201 Applied Topically for the Treatment of Hard to Heal Chronic Ulcerated Wounds
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to slow recruitment
Sponsor: Regenera Pharma Ltd (Industry)
Collaborators: TransCom Global Ltd. (CRO) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGN-WH-001
Record Dates: First submitted 2011-09-04; First posted 2011-09-07 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Chronic Wound
Keywords: chronic wound; ulcerated wound; venous insufficiency; lymphatic insufficiency; neuropathic wound; diabetic ulcer; post- operative; post-traumatic chronic wound
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: RPh201, botanical drug product

INTERVENTIONS:
Drug: RPh201, botanical drug product — topical, three times per week for a period of 4 consecutive weeks, followed by a single follow up visit 3 months post end of the last treatment day

SUMMARY:
The study objectives are to evaluate safety and efficacy of topical administration of RPh201 oil solution (botanical extract) for treatment of patients with hard to heal chronic ulcerated wounds.

DETAILED DESCRIPTION:
The study objectives are to evaluate safety and efficacy, of topical administration of RPh201 for treatment of patients with hard to heal wounds.

This is to include:

* Safety evaluation of RPh201 (botanical extract) formulated as an oil solution administered topically three times per week during an overall treatment period of up to 4 weeks in patients with hard to heal wounds.
* Efficacy assessment of wound improvement following the use of RPh201 oil solution (botanical extract) administered topically three times per week during an overall treatment period of up to 4 weeks and at the follow-up visit at 3 months after end of treatment in patients with hard to heal wounds

ELIGIBILITY:
Inclusion Criteria:

1. Participants, either men or women are ≥ 18 years of age.
2. Patients must have at least one hard to heal wound of different etiologies (venous insufficiency, lymphatic insufficiency, neuropathic wounds or diabetic ulcers, post- operative and post-traumatic chronic wounds) located on the leg shin or foot.
3. The wound is refractive to healing at least 4 weeks prior to treatment, although treated by routine practice.
4. Wound area size is in the range of: 3 - 36 square centimeters.
5. Patients defined as grade C or above on the granulometer scale (see section 6.5.1).
6. Participants understand the nature of the procedure and provide written informed consent prior to any study procedure.
7. Women of child bearing potential must use adequate birth-control precautions.

Exclusion Criteria:

1. Clinically significant arterial vascular disease with ABI index <0.45 if the peripheral pulse is not palpable, or flatted PVR in case of non palpable arteries.
2. Clinical evidence for presence of infection in the soft tissue, joint and/or bone (osteomyelitis).
3. Wound has Non-viable tissue which covers more than 50% of the wound area.
4. Patients with skin disorders unrelated to the ulcer that are presented adjacent to the wound.
5. The wound penetrates into deep organs and involves bone, tendon or joint
6. Wound with sinus tracts
7. Patients are receiving, or have received within one month prior to enrollment any treatment known to impair wound healing, including but not limited to: immuno-suppressive drugs, cytotoxic agents, radiation therapy and chemotherapy.
8. Treatment with a dressing containing growth factors or other biological dressings within 15 days, prior to the screening visit.
9. Patients that have a history of alcohol or drug abuse within the last two years.
10. Female patients who are pregnant or nursing, or of childbearing potential and are not using adequate contraception.
11. Participation in another clinical trial within 30 days prior to the Screening Visit or during this study.
12. Clinically significant and/or uncontrolled condition or other significant medical disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To determine the safety use of RPh201 administered topically three times a week during an overall treatment period of up to 4 weeks, with 52 days follow-up | 90 days
  * Safety evaluation - To demonstrate safety using the RPh201 oil solution in terms of skin irritation score to be less than 2 for erythema /edema individual subject's results or less then 1.9 for Primary Irritation Index (PII) category (see section 6.5.2 and APPENDIX 2) .
  * Safety evaluation - To demonstrate safety of using RPh201 oil solution in terms of type and severity of adverse events.

SECONDARY OUTCOMES:
To obtain preliminary data on the efficacy of RPh201 on improving wound status in patients with hard to heal chronic ulcerated wounds | 90 days
  * Evaluation of the correlation between the treatment period and changes in wound area size.
  * Assessment of wound closure state in terms of % Non-viable area, % granulation tissue appearance,
  * Assessment of wound closure state in terms of time to wound closure.
  * Assessment of pain based on a pain analog scale of 1-10.

CONTACTS AND LOCATIONS:
Overall Officials: Eran Tamir, Dr., Principal Investigator — High Risk Foot Clinic - Maccabi Health Services Tel Aviv
Locations (1):
- High Risk Foot Clinic - Maccabi Health Services, Tel Aviv, Israel